CLINICAL TRIAL: NCT07198321
Title: A Single-Arm, Open-Label, Multicenter Phase I/II Clinical Study
Brief Title: A Single-Arm, Open-Label, Multicenter Phase I/II Clinical Study of GFH276 in Patients With RAS-Mutant Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genfleet Therapeutics (Shanghai) Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GFH276X1101
Record Dates: First submitted 2025-09-15; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Cancer; PDAC; CRC (Colorectal Cancer); NSCLC
Keywords: cancer; RAS
MeSH Terms: conditions — Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GFH276 (Experimental): GFH276 will be administered at the assigned dose level, orally, until disease progression or intolerable toxicity.
  Interventions: Drug: GFH276

INTERVENTIONS:
Drug: GFH276 — GFH276 will be administered at the assigned dose level, orally, until disease progression or intolerable toxicity.

SUMMARY:
This study is an investigation to evaluate the safety/tolerability, pharmacokinetics (PK), and efficacy of GFH276 as a single agent in patients with advanced solid tumors harboring RAS mutations.

The primary objectives of the Phase I study are to assess the safety/tolerability, PK, and preliminary efficacy of GFH276 in patients with advanced solid tumors harboring RAS mutations, and to determine the Maximum Tolerated Dose (MTD) and Recommended Phase II Dose (RP2D) of GFH276.

The primary objective of the Phase II study is to evaluate the efficacy of GFH276 in patients with RAS-mutant advanced pancreatic ductal adenocarcinoma (PDAC), advanced non-small cell lung cancer (NSCLC), advanced colorectal cancer (CRC), and other advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must voluntarily agree to participate in the trial and sign a written informed consent form.
2. Male or female ≥ 18 years old and ≤75 years old.
3. ECOG performance status of 0-1.
4. With a life expectancy of ≥3 moths
5. Have at least one measurable lesion according to RECIST1.1, and the phase Ia allows no measurable lesion.
6. Adequate laboratory parameters during the screening period.

Exclusion Criteria:

1. Active brain metastases.
2. Prior treatment with a PAN-RAS inhibitor.
3. Palliative radiotherapy was completed within 14 days before the first dose.
4. Have poorly controlled or severe cardiovascular disease.
5. Subjects with active hepatitis B or active hepatitis C.
6. Known allergy to the study drug or its components.
7. Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2025-09-22 (Estimated); Primary Completion 2027-09-22 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Phase Ia:The incidence and severity of AEs and SAEs | 48 months
  The incidence and severity of AEs and SAEs
Phase Ia:The incidence of DLT events | 21 days
  The incidence of DLT events
Phase Ib:The incidence and severity of AEs and SAEs | 48 months
  The incidence and severity of AEs and SAEs
Phase II:Overall response rate (ORR) | about 48 months
  Aassessed by investigators according to RECIST 1.1
Efficacy endpoints | about 48 months
  Duration of response (DoR)

SECONDARY OUTCOMES:
Peak Plasma Concentration(Cmax) | about 48 months
DCR | about 48 months
  he percentage of patients who achieved CR, PR and SD

CONTACTS AND LOCATIONS:
Overall Officials: li zhang, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun-Yat sen university cancer center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No